CLINICAL TRIAL: NCT05183672
Title: Improving Post-acute Stroke Follow-up Care by Adopting Telecare Consultations in a Nurse-led Clinic During COVID-19 and Beyond: A Hybrid Type 2 Implementation-effectiveness Randomized Trial
Brief Title: Improving Post-acute Stroke Follow-up Care by Adopting Telecare Consultations in a Nurse-led Clinic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The Queen Elizabeth Hospital (Other)
Responsible Party: Principal Investigator, Arkers, Wong, Assistant professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: A0036516
Record Dates: First submitted 2021-12-07; First posted 2022-01-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: stroke; telecare consultation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive three tertiary stroke care consultations provided by stroke nurses via telecare in 3 months.
  Interventions: Procedure: Telecare consultation
- Control group (Placebo Comparator): Participants will receive three usual face-to-face consultations provided by stroke nurses in 3 months
  Interventions: Procedure: Usual face-to-face consultation

INTERVENTIONS:
Procedure: Telecare consultation — Using Zoom to communicate with patients
  Arms: Intervention group
Procedure: Usual face-to-face consultation — Face-to-face communication with patients
  Arms: Control group

SUMMARY:
Since 2017, Hong Kong has provided post-acute stroke services in clinics operated by stroke advanced practice nurses (APNs). Currently, the applicability of the clinics has been further limited by the emergence of the coronavirus (COVID-19) pandemic due to restrictions on visits to the clinics and tightened social distancing requirements. Telecare consultations may be a viable option for contributing more flexible, interactive, and cost-efficient care models to support stroke survivors over the longer run. The present study takes advantage of this opportunity by utilizing implementation science to simultaneously implement and evaluate a telecare model of care in a nurse-led post-acute stroke clinic.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of stroke within 1 month before enrolment, will be discharged home within a week, aged 18 or above, cognitively competent with a score equal to or greater than 22 in the Montreal Cognitive Assessment Hong Kong version, own a smartphone

Exclusion Criteria:

* have unaccompanied hearing or vision loss, cannot be reached by phone, bedbound, have no Internet connection at home, participating in other clinical trials at the same time, require physical contact, i.e. wound dressing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Chang in Degree of disability after stroke | baseline, three months when the program is completed, three months after the program is completed.
  Simplified modified Rankin scale will be used to measure the degree of disability for stroke patients. The scale has three questions to identify whether the patient has a score from 0 to 5, with higher scores representing higher degree of disability.

SECONDARY OUTCOMES:
Incidence of the recurrence of stroke | baseline, three months when the program is completed, three months after the program is completed.
  The percentage of participants who re-admitted to hospital because of recurrent stroke
Change of Quality of life, which measures an individual perception oftheir position in life. It includes physical and mental health. | baseline, three months when the program is completed, three months after the program is completed.
  Quality of life will be measured using the Hong Kong version of EuroQol 5-dimension. The scale has five subdomains, which include mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Since the scale has 5 items, each digit in the five digit codes refers to the status of each dimension, ranging from 1 for no problem, to 5 for sever problem. A higher scores indicate better quality of life.
Change of Post-stroke depression | baseline, three months when the program is completed, three months after the program is completed.
  Post-stroke depression will be measured using the Chinese version of the Geriatric Depression scale. This scale has a minimum score of 0 and a maximum score of 15. Lower scores represent lower depression level.
Change of Medication adherence | baseline, three months when the program is completed, three months after the program is completed.
  Medication adherence will be determined using the Adherence to Refills and Medications Scale. The scale produces an overall adherence score of 10-40, with lower scores indicating better adherence.
Change of Social participation | baseline, three months when the program is completed, three months after the program is completed.
  Social participation will be measured using the 11-item Reintegration to Normal Living index. This scale is used to measure whether the patient has participated in several social activities before and after occurrence of stroke. The scale yields total score from 0-22, with higher scores indicating poorer social participation.
Number of attendances at a general practitioners' office, emergency department, hospital, and general out-patient clinic | baseline, three months when the program is completed, three months after the program is completed.
  To measure the utilization of healthcare services by stroke patient before and after the intervention

OTHER OUTCOMES:
Cost effectiveness of the program | baseline, three months when the program is completed, three months after the program is completed.
  Cost and quality-adjusted life years will be collected at baseline, three months when the program is completed, and three months after the program is completed. Incremental cost-effectiveness ratios between the groups will be calculated by dividing the difference in cost by the difference in quality-adjusted life years.

CONTACTS AND LOCATIONS:
Overall Officials: Arkers Wong, Ph.D., Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Queen Elizabeth Hospital, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong AKC, Kwok VWY, Wong FKY, Tong DWK, Yuen BMK, Fong CS, Chan ST, Li WC, Zhou S, Lee AYL. Improving post-acute stroke follow-up care by adopting telecare consultations in a nurse-led clinic: Study protocol of a hybrid implementation-effectiveness trial. J Adv Nurs. 2024 Mar;80(3):1222-1231. doi: 10.1111/jan.15960. Epub 2023 Nov 10. PMID 37950400